CLINICAL TRIAL: NCT06803758
Title: Improving The Sensitivity of Teicoplanin Allergy Testing By Using Autologous Serum
Brief Title: Teicoplanin Allergy Testing Using Autologous Serum (TATAS)
Acronym: TATAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RHM CRI0456; 345535 (Other: IRAS Project ID)
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Drug Allergy
Keywords: Teicoplanin allergy testing; Autologous Serum
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Teicoplanin allergy testing using autologous serum (Other): 20 adult patients with history of anaphylaxis under anaesthesia ( the index episode), where teicoplanin has been given during the index episode will be recruited. In addition to usual skin testing with Teicoplanin directly onto the skin, we will perform skin testing with Teicoplanin- added autologous serum. The trial will be conducted as part of the same routine elective allergy skin-testing appointment for other drugs given during the index episode.
  Interventions: Diagnostic Test: Teicoplanin Allergy Testing using autologous serum

INTERVENTIONS:
Diagnostic Test: Teicoplanin Allergy Testing using autologous serum — In addition to performing teicoplanin allergy skin testing using standard recommended Teicoplanin concentration, we will perform skin testing using autologous serum, the supernatant which is obtained via centrifugation. Skin testing ( skin prick test and intradermal test) will be performed with these additional samples:
  1. STpre: Teicoplanin added to blood sample pre-centrigufation.
  2. STpost: Teicoplanin added to supernatant post-centrigufation.
  3. ST0: Supernatant with no additives ( serum negative control)

SUMMARY:
Allergy testing for Teicoplanin is much more unreliable than for other similar drugs. This means that we run the risk of missing serious Teicoplanin allergy, and these patients will be given another dose in future, not knowing that they are seriously allergic. Serious allergic reactions, also known as anaphylaxis, can be life threatening.

The patients which we recruit to our study will come to us through the perioperative allergy service. They will have had a reaction to a general anaesthetic, but will also have had teicoplanin as part of the anaesthetic.

We are not sure why allergy skin testing, which is fairly reliable for most other drugs, is so unreliable in detecting teicoplanin allergy. We do know that some drugs need to mix with proteins in the blood before they trigger an allergy. We would like to replicate this by mixing the teicoplanin with the patients' own blood and using this for the skin testing, to see if we get a more reliable result compared with the plain drug. Using the patient's own serum to do skin testing is an established test (the 'autologous serum test') used in certain immunological conditions, we are simply going to use it as a vehicle to test our theory.

We will recruit 20 adult patients referred with a recent history of anaphylaxis under anaesthesia, where teicoplanin has been given and is one of the drugs under suspicion of having caused the allergy. In addition to the usual allergy skin testing, which would be done anyway as part of standard allergy investigation, we will perform extra tests using autologous serum for this trial.

We hope to find a better way of testing for Teicoplanin allergy, so that patients are not put at risk where the allergy has been missed because of an unreliable test.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years old and above who have suffered suspected anaphylaxis under anaesthesia (the 'index episode'), where teicoplanin has been given

Exclusion Criteria:

* Patients unable to stop drugs that would interfere with skin tests prior to study- e.g. antihistamines or certain anti-psychotics
* Pregnancy
* Patients under age 18 years
* Patients with elevated baseline mast cell tryptase requiring further investigation
* Patients with blood-borne viruses such as Hep B, C and HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Does using autologous serum for skin testing yield more positive results as compared to using standard protocol of Teicoplanin Allergy skin test? | 2 years
  We will determine if testing using autologous serum for skin testing yield more positive results as compared to using standard protocol of Teicoplanin Allergy test.
  A positive skin prick test is defined as having wheals of 3x3mm or more at 15 mins. A positive intradermal test results is defined as wheal increment by 3mm in any direction after 20 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Nel, MB BCh FRCA, Study Chair — University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liccardi G, D'Amato G, Canonica GW, Salzillo A, Piccolo A, Passalacqua G. Systemic reactions from skin testing: literature review. J Investig Allergol Clin Immunol. 2006;16(2):75-8. PMID 16689179
- [Background] Savic LC, Garcez T, Hopkins PM, Harper NJ, Savic S. Teicoplanin allergy - an emerging problem in the anaesthetic allergy clinic. Br J Anaesth. 2015 Oct;115(4):595-600. doi: 10.1093/bja/aev307. PMID 26385667
- See also: Autologous serum skin test reactions in chronic spontaneous urticaria differ from heterologous cell reactions — https://pubmed.ncbi.nlm.nih.gov/33475206/
- See also: BSACI Standard Operating Procedures- Skin Prick Test — https://www.bsaci.org/guidelines/bsaci-standard-operating-procedures/
- See also: Emergency treatment of anaphylaxis — https://www.resus.org.uk/sites/default/files/2021-04/Anaphylaxis%20Summary%20Document.pdf